CLINICAL TRIAL: NCT05680012
Title: Tissue Destruction and Healing in Celiac Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Mayo Clinic (Other); California Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB22-1138; RC2DK133947 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2023-01-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Celiac Disease
Keywords: gluten-free diet; HLA-DQ2; HLA-DQ8; microbiome; metagenomics; intestinal epithelial cells
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gluten challenge group (Experimental): Diagnosis of celiac disease by intestinal biopsy and serology for at least 12 months
  Interventions: Dietary Supplement: Gluten containing snack bar
- Gluten de-challenge group (No Intervention): Suspected celiac disease either showing typical symptoms or positive celiac disease serology
- Control group (No Intervention): No history or symptoms of celiac disease

INTERVENTIONS:
Dietary Supplement: Gluten containing snack bar — Ingest snack bars containing 3 grams of gluten every day for 6 weeks.
  Arms: Gluten challenge group

SUMMARY:
The purpose of this clinical study is to learn more about celiac disease pathogenesis and clinical symptoms. In particular, this study will examine the interactions between biological factors such as, intestinal epithelial cells, microbiota, immune system, genetics, and gluten and their effect on celiac disease clinical symptoms, and severity of tissue destruction and its ability to heal in individuals with celiac disease. Information collected in the study will help researchers to generate better resources to advance celiac disease patient care.

DETAILED DESCRIPTION:
Celiac disease is an autoimmune enteropathy characterized by chronic inflammation of the small intestinal mucosa triggered by gluten uptake that occurs in genetically susceptible individuals carrying the specific class II human leucocyte antigens (HLA) DQ2 and DQ8 alleles. There is a spectrum in intestinal tissue damage associated with celiac disease. Some individuals develop inflammatory immunity in the absence of tissue damage, while others experience tissue damage ranging from partial to total villous atrophy. Persistent mucosal damage is associated with several severe complications, including lymphoproliferative malignancy and bone diseases. In addition, individuals with active celiac disease display a wide range of clinical symptoms, including metabolic defects that are not correlated to the degree of villous atrophy. Although much progress has been made in understanding celiac disease, major gaps remain in understanding biological mechanisms underlying inter-individual differences in clinical presentations and capacity to heal while maintaining a gluten-free diet.

ELIGIBILITY:
Inclusion Criteria:

Gluten challenge group:

1. Age 18 to 75 years old
2. Diagnosis of Celiac disease for at least 12 months by intestinal biopsy
3. Follow a strict gluten-free diet for at least the 12 consecutive months

Gluten de-challenge group:

1. Age 18 to 75 years old
2. Showing typical celiac disease symptoms
3. Not on a gluten-free diet

Control group:

1. Age 18 to 75 years old
2. Females who are not pregnant

Exclusion Criteria:

Gluten challenge group:

1. Diagnosis of any severe complication of celiac disease
2. Diagnosis of other chronic, active GI disease
3. Selective IgA deficiency
4. Severe reaction to gluten exposure
5. Any clinically significant diseases
6. History of significant substance or alcohol abuse
7. Pregnant or lactating
8. Diagnosis of blood clotting disorders

Gluten de-challenge group:

1. History of chronic inflammatory gastrointestinal disease
2. Gastrointestinal illness within the 4-week period prior to screening
3. History of lymphoproliferative disease
4. Uncontrolled blood clotting disorders
5. Any clinically significant diseases
6. History of significant substance or alcohol abuse

Control group:

1. Taking antibiotics, proton pump inhibitors, aspirin, or non-steroidal anti-inflammatory drugs
2. Known intestinal inflammation
3. Prior gastrointestinal surgery
4. Taking of antiplatelet agents or anticoagulants
5. Family history of celiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Gluten challenge group: quantitative analysis of intestinal villus to crypt ratios | baseline - 6 weeks
  villus to crypt ratios will be quantified on small bowel biopsy samples for the histologic quantification of intestinal responses to disease processes.
Gluten de-challenge group: quantitative analysis of intestinal villus to crypt ratios | baseline -12 months
  Villus to crypt ratios will be quantified on small bowel biopsy samples for the histologic quantification of intestinal responses to disease processes.

CONTACTS AND LOCATIONS:
Overall Officials: Bana Jabri, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - California Institute of Technology, Pasadena, California
  - The University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05680012/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05680012/ICF_001.pdf